CLINICAL TRIAL: NCT06369441
Title: Collection of Biological Specimens and Associated Health Information for Secondary Research in Future Studies
Brief Title: Collection of Biological Specimens and Associated Health Information
Status: Not yet recruiting | Type: Observational
Sponsor: Ovation.io, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Ovation-23-001
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Other Disease
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncology: Adults (aged 18 or older) who have an active cancer diagnosis with confirmatory pathology results indicating solid tumor and/or hematologic malignancy.

SUMMARY:
The purpose of this study is to collect blood samples from a large number of individuals with cancer to create a database for researchers to use in future studies. Researchers may use this database to discover new ways to detect and treat cancer and other diseases. Future studies may use stored blood samples to discover how genes affect health and disease.

ELIGIBILITY:
Inclusion Criteria:

* Are patients of participating study site clinics/clinical groups
* Are adults (aged 18 or older)
* Have an active cancer diagnosis with confirmatory pathology results indicating solid tumor and/or hematologic malignancy
* Participants may have other active diagnoses with confirmatory clinical results

Exclusion Criteria:

* Individuals who lack the capacity to provide informed consent
* Individuals known to be prisoners at time of biological specimen collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have an active cancer diagnosis with confirmatory pathology results indicating solid tumor and/or hematologic malignancy
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Biorepository | 10 years
  The objective of this study is to establish a biorepository and database of specimens to enable future research on the role of genetic factors in the biological mechanisms of diseases, including cancer, and treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Gee, PhD, Study Director — VP, Clinical Affairs, Ovation.io
Locations (1):
- Ovation.io, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes
All future research requests will be submitted to Ovation.io and reviewed to ensure that they are consistent with the permissions described in the informed consent form by Ovation.io staff. If there is a question regarding whether or not the research request is consistent with the informed consent form and Ovation.io's biorepository policies, Ovation.io will request review and approval by an appropriate IRB.
  Research teams whose study aims are in concordance with the purpose of the Ovation.io biorepository, may be granted access to specified coded datasets.In the case that a secondary research protocol requires biological specimen analysis to produce the requested dataset, Ovation.io will conduct the analysis on the relevant biological specimens stored in the biorepository and provide the results to the research team in the form of a de-identified dataset.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Biological specimens and associated data will be stored indefinitely.
Access Criteria: All expert determinations performed under this protocol will be pursuant to a business associate agreement and conducted by an individual who has the relevant education and experience to perform a health information de-identification assessment.